CLINICAL TRIAL: NCT03532490
Title: Trial of Roflumilast in Asthma Management (TRIM)
Acronym: TRIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Lung Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00156697; R34HL135361 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — Roflumilast; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast 500 mcg oral tablet (Active Comparator): 500 mcg roflumilast oral tablets will be taken every other day for the first two weeks. If participant tolerates the drug, the tablet will be taken once daily.
  Interventions: Drug: Roflumilast 500 Mcg Oral Tablet
- Placebo oral tablet (Placebo Comparator): 500 mcg placebo oral tablets will be taken every other day for the first two weeks. If participant tolerates the drug, the tablet will be taken once daily.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Roflumilast 500 Mcg Oral Tablet — The first two weeks the participant will take one tablet every other day. If well tolerated, participant will take one tablet every day.
  Other Names: Daliresp
  Arms: Roflumilast 500 mcg oral tablet
Drug: Placebo oral capsule — The first two weeks the participant will take one tablet every other day. If well tolerated, participant will take one tablet every day.
  Arms: Placebo oral tablet

SUMMARY:
There are currently no treatments to specifically target asthma in obese adults. This pilot study is being conducted to investigate how effective roflumilast is in treating asthma in participants that have a higher BMI. Roflumilast can induce weight loss, which may lead to improved asthma control.

The primary objective of TRIM is to perform a pilot placebo-controlled trial of roflumilast for the treatment of poorly controlled obese asthmatics.

DETAILED DESCRIPTION:
TRIM is a 24 week, randomized, double-masked, placebo controlled trial that will enroll 38 participants.

This study will be take place in seven centers of the American Lung Association- Airways Clinical Research Centers (ALA-ACRC). The centers include: Northwestern University Feinberg School of Medicine, Mount Sinai Icahn School of Medicine, Duke University, University of Arizona, the University of Vermont, The University of Alabama Lung Health Center, and University of Illinois Breathe Chicago Center. Johns Hopkins University will be the Data Coordinating Center (DCC) for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma on regular prescribed controller therapy for at least 3 months
* Previous (within five years) evidence of at least a 12% increase in forced expiratory volume at one second FEV1 after inhaling 2-4 puffs of albuterol or a positive methacholine challenge or patient reported history of improvement of asthma exacerbation after a course of systemic or inhaled corticosteroids
* Age: ≥18 years of age
* Obese: Body Mass Index (BMI) > 30 kg/m2
* Poorly controlled asthma: Asthma Control Test (ACT) Score < 20, or use of rescue inhaler, on an average of> 2 uses/week for preceding month, or nocturnal asthma awakening, on an average of 1 or more times / week in preceding month, or emergency department (ED)/hospital visit or prednisone course for asthma in past six months.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Participation in an investigational study within the past 4 weeks
* Physician diagnosis of chronic obstructive pulmonary disease
* Any condition that puts the participant at risk from weight loss as judged by the site physician
* Liver cirrhosis
* Major psychiatric disorders such as generalized anxiety disorder, major depressive disorder, history of suicidal ideation/ attempt, panic disorder, post-traumatic stress disorder, schizophrenia, schizoaffective, substance abuse or other disorders that in the opinion of the study physician that would affect study participation
* > 0 time use of illicit drugs in the past 12 months
* > 0 time use of cannabis in the past 12 months
* Uncontrolled depression as defined by a score of 15 or greater on the depression questions of the Patient Health Questionnaire (PHQ-9)
* Suicidal ideation (a score of greater than 0 on Question 9 on the PHQ-9)
* Uncontrolled anxiety as defined by a score of 10 or greater on the anxiety questions of the Generalized Anxiety Disorder 7-item (GAD-7)
* Pregnancy/lactation
* Females of childbearing age who do not agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.
* Greater than 20 pack year smoking history, or smoking within the last 6 months.
* History of bariatric surgery
* Drugs metabolized by cytochrome P450 (rifampicin, phenobarbital, carbamazepine, phenytoin, erythromycin, ketoconazole, cimetidine, fluvoxamine, enoxacin, oral contraceptives containing ethinyl estradiol with gestodene).
* Currently on roflumilast or theophylline (patient may wash out of these medications for 4 weeks prior to visit 1)
* Intention to move out of area within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dixon, MD, Principal Investigator — University of Vermont; Robert Wise, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (7):
- United States (7):
  - University of Alabama Lung Health Center, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Illinois at Chicago, Breathe Chicago Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mount Sinai Icahn School of Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - University of Vermont, Colchester, Vermont

REFERENCES:
- [Derived] Dixon AE, Que LG, Kalhan R, Dransfield MT, Rogers L, Gerald LB, Kraft M, Krishnan JA, Johnson O, Hazucha H, Roy G, Holbrook JT, Wise RA. Roflumilast May Increase Risk of Exacerbations When Used to Treat Poorly Controlled Asthma in People with Obesity. Ann Am Thorac Soc. 2023 Feb;20(2):206-214. doi: 10.1513/AnnalsATS.202204-368OC. PMID 36170654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2018 and last participant visit was completed on July 2021. Participants were recruited from 7 clinical sites: University of Vermont, University of Arizona, Duke, University of Illinois, Chicago, Northwestern, University of Alabama, and Mount Sinai.
Period: Overall Study
Arm/Group | Placebo Oral Tablet | Roflumilast 500 mcg Oral Tablet
Started | 16 | 22
Completed | 16 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Tablet | Roflumilast 500 mcg Oral Tablet | Total
Number analyzed (Participants) | 16 | 22 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [50 to 63] | 51 [43 to 59] | 53 [49 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 14 | 19 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 22 | 38
Smoking status [Count of Participants; unit: Participants]
  Never | 14 | 18 | 32
  Former | 2 | 4 | 6
Age at asthma onset (years) [Median (Inter-Quartile Range); unit: years] | 14 [9 to 37] | 21 [7 to 42] | 21 [7 to 42]
Asthma Control Test at Visit 2 (V2) [Median (Inter-Quartile Range); unit: units on a scale] — Range 5-25, higher score is indicative of better health
  units on a scale | 19 [16 to 19] | 17 [14 to 18] | 17 [15 to 19]
Asthma Symptom Utility Index [Median (Inter-Quartile Range); unit: units on a scale] — range 0-1, higher score is indicative of better health
  units on a scale | .8 [.7 to .9] | .7 [.6 to .8] | .7 [.6 to .8]
Marks Asthma Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — Range 1-4, lower score is indicative of better health
  units on a scale | 2.1 [1 to 4] | 1.8 [1.6 to 2.4] | 2 [1.5 to 2.5]
Patient Health Questionnaire-9 [Median (Inter-Quartile Range); unit: units on a scale] — range 0-27, lower score is indicative of better health
  units on a scale | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 4]
General Anxiety Disorder-7 [Median (Inter-Quartile Range); unit: units on a scale] — range 0-27, lower score is indicative of better health
  units on a scale | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 1]
Short form survey-36 [Median (Inter-Quartile Range); unit: units on a scale] — Range 0-100, higher score is indicative of better health
  units on a scale | 59 [46 to 76] | 67 [52 to 78] | 62 [47 to 78]
Gastrointestinal Symptom Rating Scale [Median (Inter-Quartile Range); unit: units on a scale] — range 1-7, lower score is indicative of better health
  units on a scale | 1.4 [1.2 to 2.1] | 1.5 [1.1 to 1.9] | 1.4 [1.1 to 1.9]
Forced expiratory volume at one second [Median (Inter-Quartile Range); unit: liters] | 1.91 [1.27 to 2.25] | 2.17 [1.79 to 2.41] | 2.03 [1.65 to 2.31]
Forced Vital Capacity [Median (Inter-Quartile Range); unit: liters] | 3 [2.55 to 3.23] | 3.08 [2.75 to 3.52] | 3.08 [2.75 to 3.23]
Forced Expiratory Volume/Forced vital capacity [Median (Inter-Quartile Range); unit: ratio] | .78 [.70 to .83] | .76 [.69 to .78] | .76 [.70 to .81]
Methacholine PD20 [Median (Inter-Quartile Range); unit: microgram (mcg)] | 115 [14 to 236] | 75 [37 to 162] | 95 [14 to 236]
Greater than/equal to 1 unscheduled health visit for asthma in prior year [Count of Participants; unit: Participants] | 10 | 8 | 18
Greater than/equal to 1 course of oral corticosteroids in prior year [Count of Participants; unit: Participants] | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Test Score
Description: The Asthma Control Test was designed to help participants describe their asthma and how it affects how they feel and what they are able to do. They choose a response based on their asthma within the last 4 weeks. Participants select how many times per week they experience different asthma symptoms and how often they had to use a rescue inhaler or nebulizer. There are 5 questions with 5 responses; 1 meaning their asthma is not well controlled or they had symptoms more frequently, through 5 meaning they feel their asthma is well controlled or they do not experience any symptoms.
  The primary outcome is an unadjusted comparison of 24 week change in Asthma Control Test scores between the treatment groups.
Time Frame: Baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Placebo: 500 mcg placebo oral tablets will be taken every other day for the first two weeks. If participant tolerates the drug, the tablet will be taken once daily.
  Placebo oral capsule: The first two weeks the participant will take one tablet every other day. If well tolerated, participant will take one tablet every day.
- Roflumilast: 500 mcg roflumilast oral tablets will be taken every other day for the first two weeks. If participant tolerates the drug, the tablet will be taken once daily.
  Roflumilast 500 Mcg Oral Tablet: The first two weeks the participant will take one tablet every other day. If well tolerated, participant will take one tablet every day
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on a scale | 2 [.7 to 3.3] | 2.6 [.5 to 4.4]

2. Secondary Outcome: Change in Weight
Description: Weight change measured in kilograms (kg).
Time Frame: Baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Placebo Oral Tablet | Roflumilast 500 mcg Oral Tablet
Number analyzed (Participants) | 16 | 22
kg | -1.7 [-2.9 to -0.5] | -2.2 [-4.2 to -0.1]

3. Secondary Outcome: Change in Asthma Symptom Utility Index (ASUI)
Description: A 10-item questionnaire, patient preference-based scale assessing frequency and severity of selected asthma-related symptoms and treatment side effects, for use in clinical trials and cost-effectiveness studies in asthma. Range is 0-1. Higher score is indicative of better health.
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on a scale | .14 [.07 to .21] | .16 [.09 to .23]

4. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS)
Description: It has 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). Subscale scores range from 1 to 7 and higher scores represent more discomfort and poor health.
Time Frame: Baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on scale | -.1 [-.4 to .2] | 0.0 [-.3 to .2]

5. Secondary Outcome: Change in Generalized Anxiety Disease (GAD-7)
Description: GAD-7 has 7 questions. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. The following cut-offs correlate with level of anxiety severity:
  Score 0-4: Minimal Anxiety Score 5-9: Mild Anxiety Score 10-14: Moderate Anxiety Score greater than 15: Severe Anxiety
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on scale | 0.0 [-.5 to .5] | 0.0 [-.8 to .6]

6. Secondary Outcome: Change in Marks Asthma Quality of Life Questionnaire
Description: 20 items with 2 week recall. Self-administered questionnaire intended for use with adults. Respondents are asked to describe how troubling particular items have been over the past four weeks. Covers both physical and emotional impact. Range 1-4. lower score is indicative of better health
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on scale | -.3 [-.6 to 0.0] | -.4 [-.6 to -.25]

7. Secondary Outcome: Change in SF 36
Description: The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. Range 0-100. Higher score is indicative of better health.
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on scale | 6.4 [2.8 to 10.0] | 5.5 [2.5 to 8.6]

8. Secondary Outcome: Change in PHQ9
Description: The PHQ-9 (Patient Health Questionnaire-9) objectifies and assesses degree of depression severity via questionnaire. It has 9 questions. Range 0-27, lower score is indicate of better health.
Time Frame: baseline and 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on scale
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 16 | 22
units on scale | -.6 [-1.6 to .5] | 0.0 [-.8 to .8]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo Oral Tablet | Roflumilast 500 mcg Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/16 | 6/22
Other Adverse Events (participants affected / at risk) | 10/16 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Tablet (N=16) | Roflumilast 500 mcg Oral Tablet (N=22)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Loss of appetite (General disorders) | 0 (0) | 2 (2)
Dehydration (General disorders) | 0 (0) | 1 (1)
Abdominal pain (umbilical hernia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Tablet (N=16) | Roflumilast 500 mcg Oral Tablet (N=22)
Headache (General disorders) | 0 (0) | 7 (7) — Treatment emergent
Congestion, runny nose, sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) — Treatment emergent
Acute upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — Treatment emergent
Chest discomfort (Cardiac disorders) | 0 (0) | 2 (2)
chest pain (Cardiac disorders) | 0 (0) | 2 (2) — Treatment emergent
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) — Treatment emergent
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — Treatment emergent
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Treatment emergent
Skin rash (General disorders) | 1 (1) | 2 (2) — Treatment emergent
Muscle pain/aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Treatment emergent
Any emergent symptoms (General disorders) | 4 (4) | 13 (13) — Treatment emergent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03532490/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03532490/ICF_003.pdf